CLINICAL TRIAL: NCT04338555
Title: Effects of Transcutanclus Electrical Acupoint Stimulation on Postoperative Cognitive Dysfunction in Elderly Patients
Brief Title: Effects of TEAS on POCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Jie Tian, Dr., RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AES20200407
Record Dates: First submitted 2020-04-06; First posted 2020-04-08 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Post-operative Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEAS group (Experimental): Patients in the TEAS group will receive electrical stimulation of acupoints at Neiguan and Shenmen points for 30min every hour. The stimulation will repeat until the end of surgery.
  Interventions: Procedure: Transcutaneous electrical acupoint stimulation
- control group (No Intervention): In patients from the control group, the electrodes will only be attached to the corresponding sites, with no TEAS electrical stimulation given during the operation.

INTERVENTIONS:
Procedure: Transcutaneous electrical acupoint stimulation — TEAS group will receive electrical stimulation of acupoints at Neiguan and Shenmen points for 30 min every hour during the surgery.
  Arms: TEAS group

SUMMARY:
Patients undergoing elective orthopedics, urology, and general surgery will be included and randomly allocated to TEAS group or control group . After routine anesthesia induction and tracheal intubation, patients in TEAS group will receive electrical stimulation of acupoints at Neiguan and Shenmen points. For patients in the control group, the electrodes will be only attached to the corresponding sites, with no TEAS electrical stimulation given during the operation. The primary outcome is the incidence of POCD at Day 7 after surgery. The secondary outcomes include the incidence of POD during post-operative days 1-7, the incidence of POCD at Day 30 after surgery, and the serum levels of cytokines, including IL-1β、IL-6、TNF-α、MMP9 on Day 1 after surgery.

DETAILED DESCRIPTION:
This study will enroll 110 patients who are older than 60 years old and will have elective orthopedics, urology, or general surgeries under general anesthesia. Patients will be randomly assigned to TEAS group and control group. After routine anesthesia induction and tracheal intubation, patients in TEAS group will receive electrical stimulation of acupoints at Neiguan and Shenmen points for 30min every hour. In other words, the patients will receive TEAS stimulation for 30min, then no stimulation for 30min, then stimulation for another 30min, etc, until the end of the surgery. For patients in the control group, the electrodes will be only attached to the corresponding sites, with no TEAS electrical stimulation given during the operation. The primary outcome is the incidence of POCD at Day 7 after surgery. The secondary outcomes include the incidence of POD during post-operative days 1-7, the incidence of POCD at Day 30 after surgery, and the serum levels of cytokines, including IL-1β、IL-6、TNF-α、MMP9 on Day 1 after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. ≧ 60 years old;
2. communicate normally；
3. ASA Physical Status 1-2;
4. Patients will have elective orthopedics, urology or general surgeries under general anesthesia;
5. With an estimated surgery time of more than 2h;
6. Agree to participate the trial.

Exclusion Criteria:

1. Patients with brain diseases or history of brain diseases;
2. Preoperative diagnosis of cognitive impairment by subtle mental state (MMSE) less than 24 points;
3. Patients with history of neurological and psychological disorders including AD, stroke, and psychosis;
4. Severe hearing or visual impairment, illiteracy;
5. preoperative systolic blood pressure >190mmHg, or diastolic blood pressure >100mmHg;
6. Disagree to participate in this research;
7. Have used other medical electronic devices.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
the incidence of POCD | at Day 7 post-surgery
  cognitive function of the patients will be analyzed with MMSE, Digital breadth, Number symbol, Visual regeneration, Color word conversion, Color Trail Marking Test (PartB) and CAM, and reflected by Z score with the following formula: Z=（Xafter-Xbefore）/SDbefore

SECONDARY OUTCOMES:
the incidence of POCD | at Day 30 post-surgery
  cognitive function of the patients will be analyzed with MMSE, Digital breadth, Number symbol, Visual regeneration, Color word conversion, Color Trail Marking Test (PartB) and CAM, and reflected by Z score with the following formula: Z=（Xafter-Xbefore）/SDbefore
the incidence of delirium | from Day 1 to Day 7 post-surgery
  whether the patients develop delirium will be analyzed with CAM
serum IL-1β level | at Day 1 post-surgery
  an inflammatory mediator that reflects systemic inflammation
serum IL-6 level | at Day 1 post-surgery
  an inflammatory mediator that reflects systemic inflammation
serum TNF-α level | at Day 1 post-surgery
  an inflammatory mediator that reflects systemic inflammation
serum MMP9 level | at Day 1 post-surgery
  an inflammatory mediator that reflects systemic inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Jie Tian, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, China